CLINICAL TRIAL: NCT02241525
Title: Individually Optimized Uniform Contrast Enhancement in CT Angiography for the Diagnosis of Pulmonary Thromboembolic Disease
Brief Title: CT for Pulmonary Thromboembolic Disease
Acronym: CT for PE
Status: Terminated | Type: Observational
Why Stopped: The PI left the university
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Site Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00063432
Record Dates: First submitted 2014-08-29; First posted 2014-09-16 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary; Thromboembolic; Lung
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective: Twenty patients will be enrolled and scanned with the RESEARCH procedures
- Retrospective: Patients with matching age and BMI will be selected from existing patients with a CLINICAL STANDARD of Care CTPA scan.

SUMMARY:
Examine the feasibility and efficacy of individually optimized uniform contrast enhancement in CT pulmonary angiography (CTPA) for the diagnosis of pulmonary thromboembolic disease.

DETAILED DESCRIPTION:
Patient characteristics, qualitative image quality scores, and quantitative contrast enhancement and CNR will be described using mean values and standard deviations for continuous variables, and frequencies and percent for categorical variables. Difference between the two patient groups will be compared using Wilcoxon signed rank tests and chi-square statistics for continuous and categorical variables, respectively. All statistical tests will be performed at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patients who have been recommended for CTPA scan for the diagnosis of pulmonary; thromboembolic disease (PE) in the Department of Diagnostic Radiology and Nuclear Medicine at the University of Maryland-Patients whose body mass index (BMI) is greater than 30 kg/m2.
* Patients whose body mass index (BMI) is greater than 30 kg/m2
* Patients who signed the University of Maryland Medical Center Consent for Intravenous Contrast Administration

Exclusion Criteria:

* Pregnant or breast-feeding women; Female participants of childbearing age (10 - 60 years) will be screened for their pregnancy status prior to study registration, by following the Department of Diagnostic Radiology and Nuclear Medicine CLINICAL STANDARD Procedure DI-AOP-003 "Pregnancy Screening Documentation"; - Patients with decreased renal function34-36. This is evaluated by blood work checked within 30 days prior to the CTPA scan with contrast. Patients cannot receive contrast if their BUN index is not within [7-20] or creatinine is not within [0.5 - 1.4] mg/dL
* Patients with decreased renal function34-36. This is evaluated by blood work checked within current admission for inpatients or within 30 days for outpatients prior to the CTPA scan with contrast. Patients cannot receive contrast if their serum creatinine level exceeds 2.0 mg/dL
* Patients with known moderate or severe allergic reactions to contrast, including but not limited to: shortness of breath, a change in baseline vital signs, such as a change in blood pressure, tachycardia, increased respirations that can progress to major respiratory distress, laryngeal edema, bronchospasm, arrhythmias, convulsions, and cardiopulmonary arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients for a diagnosis of PE
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of patients with individually optimized bi-phasic contrast injection for CTPA scan | 1 year
  The primary endpoint is to study the feasibility( bi-phasic vs. singular pahse contrast injection (by comparison analysis)) of individually optimized bi-phasic contrast injection for CTPA scan.
Efficacy of PE diagnosis with CTPA imaging | 1 year
  To quantify the efficacy (by comparison analysis) of PE diagnosis of this new contrast injection protocol in terms of reduced frequency of non-diagnostic CTPA image vs. standard of care procedures.

SECONDARY OUTCOMES:
# of patients who receive contrast enhancement and CNR of CTPA scans | 1 year
  A secondary endpoint is to quantitatively evaluate (by comparison analysis) the contrast enhancement and CNR of CTPA scans. Twenty patients (20) will be enrolled and scanned with the RESEARCH procedures. Another twenty retrospective patients (20) with matching age and BMI will be selected from existing patients with a CLINICAL STANDARD of Care CTPA scan and enrolled on retrospective protocol:
  HP-00056512 "Individually optimized uniform contrast enhancement in CT angiography for the diagnosis of pulmonarythromboembolic disease - A simulation study".

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, PhD, Principal Investigator — Univerysity of Maryland Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No